CLINICAL TRIAL: NCT04769258
Title: Effectiveness and Safety of COVID-19 Vaccine in Patients With Inflammatory Bowel Disease Treated With Immunomodulatory or Biological Drugs
Brief Title: Effectiveness and Safety of COVID-19 Vaccine in Patients With IBD Treated With Immunomodulatory or Biological Drugs (ESCAPE-IBD)
Acronym: ESCAPE-IBD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Italian Group for the study of Inflammatory Bowel Disease (IG-IBD) (Other)
Responsible Party: Sponsor
Other Study IDs: IGIBD001
Record Dates: First submitted 2021-02-04; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — 2019-nCoV Vaccine mRNA-1273; ChAdOx1 nCoV-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with IBD treated with immunomodulatory drugs
  Interventions: Biological: Pfizer Comirnaty vaccine
- Patients with IBD not treated with the immunomodulatory drugs
  Interventions: Biological: Pfizer Comirnaty vaccine

INTERVENTIONS:
Biological: Pfizer Comirnaty vaccine — COVID 19 vaccines administered to the patients according to the times and modalities established by the Italian National Vaccination Plan. Further vaccines will be evaluated if and when they are available in Italy during the study period.
  Other Names: Moderna (Moderna vaccine, mRNA-1273); Astrazeneca (Oxford-Astrazeneca, ChAdOx1)

SUMMARY:
The COVID-19 pandemic has led to initial concerns for patients with Inflammatory Bowel Disease treated with immunosuppressive drugs, as they could be theoretically exposed to a higher risk of SARS-CoV-2 infection and/or severe forms of COVID-19.

Although initial studies have not shown an increased risk of developing SARS-CoV-2 disease related to immunosuppressive therapy, robust data are not yet available to allow for risk stratification. In this regard, the availability of vaccines represents a cornerstone in the management of the pandemic. Unfortunately, patients on immunosuppressive drugs have largely been excluded from the trials of COVID-19 vaccines, creating potential concerns regarding the validity of their efficacy for IBD patients treated with immunosuppressive agents.

DETAILED DESCRIPTION:
This is a 12-month, prospective, multicentre, case-control, observational study comparing effectiveness and safety of COVID-19 vaccine in patients with IBD treated with immunomodulatory drugs (cases) compared with those not treated with the aforementioned drugs (controls). The study should be regarded as observational because the participants will receive the intervention (Covid-19 Vaccine) as part of routine medical care (the administration will be performed outside the study and according to the times and modalities established by the Italian National Vaccination for the whole Italian population aged 18 and over). Then, we aim to assess the effect of this intervention in two predefined groups of individuals (cases and controls). All consecutive patients admitted at each IG-IBD centre that agree to participate in this study could be screened for inclusion. In case of patient's refusal to COVID-19 vaccination, this will be recorded in order to estimate the rate of adherence to the vaccination. Similarly, patients willing to vaccinate but unable to participate in the study due to logistic problems (for example; long distance from the IBD centre) will be recorded.

After enrollment, each patient will be visited at baseline; the interval between basal visit and the subsequent vaccine shall not exceed 10 days. The vaccine will be administered to the patients according to the times and modalities established by the Italian National Vaccination Plan. After the last dose of the vaccine, each patient will enter a 12 month follow-up period. An additional follow-up period will be admitted, as required by clinicians, in order to further evaluate ongoing adverse events.

At baseline, all enrolled patients will undergo a detailed assessment including: demographics, smoking status, body mass index, co-morbidities (presence of diabetes, arterial hypertension, chronic obstructive pulmonary disease, heart disease, and so on), stratification of the disease according to the Montreal classification, activity of the disease (assessed with Harvey-Bradshaw Index for CD, and Partial Mayo Score for UC), current medications, laboratory parameters (haemoglobin, white blood cells, C-reactive protein, faecal calprotectin). Furthermore, all enrolled patients will be tested for the quantitative detection of IgM and IgG antibodies against SARS-CoV-2. In case of IgM positivity, patients will be invited to perform a nasopharyngeal swab for the detection of SARS-CoV-2 RNA. The safety of the vaccine will be assessed by considering the incidence of reported adverse events, which will be reported by the patients during the 10 days following the administration of the vaccine (single assessment in case of single-dose vaccine, double assessment in case of double-dose vaccines, i.e. one evaluation for each dose). After 2 and 12 months from the last dose of the vaccination, the quantitative detection of IgM/IgG antibodies against SARS-CoV-2 will be repeated. The dosage of antibodies will be centrally performed at IEO in Milan. In addition, a proactive surveillance will be performed at 3,6, and 12 months - preferably combined with pre-scheduled direct visits, or alternatively via remote contacts - to detect new or suspected diagnosis of COVID-19. In case of active symptoms suspected for COVID-19 without an established diagnosis, patients will be invited to perform a nasopharyngeal swab for the detection of SARS-CoV-2 RNA. The proactive surveillance will also involve the occurrence of adverse events to the vaccine and the assessment of disease activity to detect flare-ups of IBD (see timeline).

All data will be collected anonymously in a specifically arranged eCRF form inside the IG-IBD registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, without racial restriction, aged 18 years or older, willing to receive the COVID-19 vaccine
* An established diagnosis of Crohn's disease or Ulcerative Colitis or unclassified colitis
* Current treatment with conventional immunosuppressants (steroids, azathioprine, 6-mercaptopurine, methotrexate), biologics (infliximab, adalimumab, golimumab, vedolizumab, ustekinumab), or small molecule drugs (tofacitinib): will be included as cases
* Currently off-therapy or treated with mesalamine only: will be included as controls
* Capability to express a written informed consent for COVID-19 vaccination
* Capability to express a written informed consent for the study

Exclusion Criteria:

* Primary immunodeficiencies and human immunodeficiency virus infection

  * Vaccination against SARS-CoV-2 already performed before enrolment
  * Contraindications to COVID-19 vaccine or intolerance to its components
  * Documented history of previous occurrence of COVID-19
  * Documented history of previous occurrence of asymptomatic SARS-CoV2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 690 patients with IBD treated with immunomodulatory drugs (cases) and 690 patients with IBD not treated withimmunomodulatory drugs (controls)
Sampling Method: Probability Sample
Enrollment: 1380 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative serum titer of IgM and IgG against SARS-CoV-2 | 12 months from the vaccination
  To evaluate the quantitative serum titer of IgM and IgG against SARS-CoV-2 after 2 and 12 months from the vaccination in patients with IBD treated with conventional immunosuppressants, biologics, or small molecule drugs (cases) compared with IBD patients not treated with the aforementioned drugs (i.e. off-therapy, or treated with mesalamine only - controls).

SECONDARY OUTCOMES:
Rate of COVID-19 occurrence | 12 months from the vaccination
  To assess the rate of COVID-19 occurrence over a temporal end-point of one year from the last dose of the vaccination
Rate of adherence to the vaccination | 12 months from the vaccination
  To assess the rate of adherence to the vaccination by identifying the patients not willing to be vaccinated during screening
Rate of adverse events of the different vaccines | 12 months from the vaccination
  To assess the rate of adverse events of the different vaccines
Rate of IBD flare-ups | 12 months from the vaccination
  To assess the rate of IBD flare-ups occurring within 3 months from the last dose of vaccine to those occurring thereafter
Predictors of effectiveness of COVID-19 vaccine | 12 months from the vaccination
  To assess the predictors of effectiveness of COVID-19 vaccine at baseline.in terms of quantitative serum titer of IgM and IgG against SARS-CoV-2 after 2 and 12 months from the vaccination (primary objective) and of the rate of COVID-19 occurrence over a temporal end-point of one year from the last dose of the vaccination (one of the secondary objectives).
Differences of effectiveness between patients | 12 months from the vaccination
  To detect differences of effectiveness between patients treated with different immunomodulators.in terms of quantitative serum titer of IgM and IgG against SARS-CoV-2 after 2 and 12 months from the vaccination (primary objective) and of the rate of COVID-19 occurrence over a temporal end-point of one year from the last dose of the vaccination (one of the secondary objectives).
Differences of effectiveness between the several vaccines | 12 months from the vaccination
  To detect differences of effectiveness between the several vaccines that will be available.in terms of quantitative serum titer of IgM and IgG against SARS-CoV-2 after 2 and 12 months from the vaccination (primary objective) and of the rate of COVID-19 occurrence over a temporal end-point of one year from the last dose of the vaccination (one of the secondary objectives).

REFERENCES:
- [Derived] Principi M, Macaluso FS, Todeschini A, Facciotti F, Contaldo A, Castiglione F, Nardone OM, Spagnuolo R, Doldo P, Riguccio G, Conforti FS, Vigano C, Ascolani M, Fiorino G, Correale C, Bodini G, Milla M, Scardino G, Vernero M, Desideri F, Caprioli F, Mannino M, Rizzo G, Orlando A; Italian Group for the study of Inflammatory Bowel Disease (IG-IBD). Safety, hesitancy of coronavirus disease 2019 vaccination and pandemic burden in patients with inflammatory bowel disease: data of a national study (ESCAPE-IBD). Eur J Gastroenterol Hepatol. 2023 Jun 1;35(6):629-634. doi: 10.1097/MEG.0000000000002550. Epub 2023 Apr 4. PMID 37115976
- [Derived] Macaluso FS, Principi M, Facciotti F, Contaldo A, Todeschini A, Saibeni S, Bezzio C, Castiglione F, Nardone OM, Spagnuolo R, Fantini MC, Riguccio G, Caprioli F, Vigano C, Felice C, Fiorino G, Correale C, Bodini G, Milla M, Scardino G, Vernero M, Desideri F, Mannino M, Rizzo G, Orlando A; Italian Group for the study of Inflammatory Bowel Disease (IG-IBD). Reduced humoral response to two doses of COVID-19 vaccine in patients with inflammatory bowel disease: Data from ESCAPE-IBD, an IG-IBD study. Dig Liver Dis. 2023 Feb;55(2):154-159. doi: 10.1016/j.dld.2022.08.027. Epub 2022 Aug 29. PMID 36127228